CLINICAL TRIAL: NCT04696900
Title: Examination of the Effect of Prescribed Cardiac Rehabilitation on Quality of Life, Exercise Capacity and Course of Disease in Patients With Advanced Heart Failure or After Ventricular Assist Device Implantation
Brief Title: Effect of Prescribed Cardiac Rehabilitation in Patients With Advanced Heart Failure or Ventricular Assist Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REHAB-HF/VAD
Record Dates: First submitted 2020-02-04; First posted 2021-01-06 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
Keywords: advanced heart failure; ventricular assist device; exercise training; cardiac rehabilitation
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise training (Other): 14 participants will absolve a prescribed exercise training for 12 months.
  Interventions: Procedure: Exercise training

INTERVENTIONS:
Procedure: Exercise training — exercise training in an approved rehabilitation program

SUMMARY:
This trial will evaluate the effect of prescribed exercise training on quality of life and exercise capacity of patients with advanced heart failure or after ventricular assist device implantation. Furthermore, clinical, laboratory and echocardiographic markers of heart failure, rehospitalization rates and cost-effectiveness will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age >17 years
* written informed consent
* chronic end-stage systolic heart failure with or without ventricular assist device
* clinically stable for at least 6 weeks
* prescription of cardiac rehabilitation

Exclusion Criteria:

* addictions or other illnesses that impact the ability to understand the nature, scope and consequences of the trial
* lack of knowledge of German to fully understand study information
* pregnancy, pre-menopausal women
* participation in the rehabilitation program < 80%
* contraindications of cardiopulmonary exercise testing on an ergometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of exercise training in severe heart failure as assessed by quality of life | after 3, 6 and 12 months
  Change of quality of life by Kansas City Cardiomyopathy Questionnaire
Efficacy of exercise training in severe heart failure as assessed by exercise capacity | after 3, 6 and 12 months
  Change of exercise capacity measured by six-minute walking distance in meters

SECONDARY OUTCOMES:
rehospitalization rates | 12 months before training and 12 months while training
  Change in rehospitalization rate or unplanned outpatient healthcare visits due to symptoms of heart failure measured by a final visit and record screening
heart failure biomarkers | after 6 and 12 months
  Change in biomarkers of heart failure: NTproBNP
Renal function biomarker: Creatinin | after 6 and 12 months
  Change in biomarkers of renal function: creatinin
Renal function biomarkers: glomerular Filtration rate | after 6 and 12 months
  Change in biomarkers of renal function: glomerular filtration rate
Hepatic function biomarkers: transaminases | after 6 and 12 months
  Change in biomarkers of hepatic function: transaminases
Hepatic function biomarkers: gamma-glutamyltransferase | after 6 and 12 months
  Change in biomarkers of hepatic function: gamma-glutamyltransferase
Heart failure Progression: Ejection fractions | after 6 and 12 months
  Change of echocardiographic findings: ejection fraction (in %)
Heart failure Progression: Diameters | after 6 and 12 months
  Change of echocardiographic findings: diameters (in mm)
Heart failure Progression: Aortic Valve opening | after 6 and 12 months
  Change of echocardiographic findings: aortic valve opening
Heart failure Progression: Valvular regurgitations | after 6 and 12 months
  Change of echocardiographic findings: Valvular regurgitation (in grades I-III°)

CONTACTS AND LOCATIONS:
Overall Officials: I A Just, Principal Investigator — German Heart Institute; F Schoenrath, Principal Investigator — German Heart Institute
Locations (1):
- German Heart Institute, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No